CLINICAL TRIAL: NCT03966508
Title: Test-retest Reliability of Measuring the Area and Intensity of Secondary Hyperalgesia Induced by High Frequency Stimulation of Skin Nociceptors
Brief Title: Reliability of Measuring the Area and Intensity of Secondary Hyperalgesia Induced by High Frequency Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HFS reliability
Record Dates: First submitted 2019-04-30; First posted 2019-05-29 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-04

CONDITIONS: Hyperalgesia, Secondary
Keywords: central sensitization; High-frequency electrical stimulation
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hyperalgesia measurement (Experimental)
  Interventions: Procedure: High-frequency electrical stimulation

INTERVENTIONS:
Procedure: High-frequency electrical stimulation — High-frequency stimulation will be applied on the volar forearm (6-10 cm distal to the cubital fossa). To avoid any confounding effect of handedness, the arm onto which HFS will be applied twice (dominant vs nondominant) will be counterbalanced across participants. HFS will consist of 12 trains of 42 Hz electrical pulses lasting 1 s each. The time interval between each train will be 10 s. The intensity of stimulation will be 5mA. Electrical pulses will be delivered to the skin using a specifically-designed electrode designed: the cathode consists of 16 blunt stainless-steel pins with a diameter of 0.2 mm protruding 1 mm from the base. The 16 pins are placed in a circle with a diameter of 10 mm. The anode consists of a surrounding stainless-steel ring having an inner diameter of 22 mm and an outer diameter of 40 mm. This procedure induces secondary pinprick hyperalgesia (an increase in pinprick sensitivity in a large area of the skin).

SUMMARY:
This study is designed to evaluate the method of assessing the and intensity areas of secondary hyperalgesia induced by High Frequency Stimulation (HFS). Measures of the areas of secondary hyperalgesia will take place on two experimental days separated by a minimum of two weeks. Each experimental day, the areas of secondary hyperalgesia will be assessed three times, starting 30 minutes following HFS. Furthermore, the investigators will assess if anxiety, catastrophization, stress and demographic variables modulate the extend of hyperalgesia.

DETAILED DESCRIPTION:
This prospective cohort study is designed to evaluate the method of assessing the areas and intensity of secondary hyperalgesia following High Frequency Stimulation (HFS), and will consist of two experimental days separated by a minimum of two weeks. During the two each session (Day1 and Day2), subjects will go through the HFS procedure on the same forearm. Then, after a 30 minutes break, the area and intensity of secondary hyperalgesia induced by HFS will be assessed three times (Time9-14), with a two-minute break between each assessment.

Before the experiment, subjects will fill two questionnaires by email : the Spielberger Trait anxiety inventory and the Pain catastrophization scale.The first experimental day, the patients will be seated on a chair and informed consent will be gained. Subjects will provide demographic information to the researcher (age, gender, size) (Time1). Then, the forearm skin of the selected arm will be marked with a pen to improve the precision of subsequent measures. The subject will then observe a period of rest for 5 minutes, to provide a baseline measure of heart rate variability.

Next, the patients will be asked to rate the pain induced by pin-prick stimulation in the area surrounding the electrode (Time2).

Following standardized explanation of the HFS procedure, the subject will fill the Spielberger State anxiety inventory (Time5), and HFS will be applied on the volar forearm (6-10 cm distal to the cubital fossa) (Time6). To avoid any confounding effect of handedness, the arm onto which HFS will be applied (dominant vs nondominant) will be counterbalanced across participants. In summary, HFS will consist of 12 trains of 42 Hz electrical pulses (pulse width: 2 ms) lasting 1 s each. The time interval between each train will 10 s. The intensity of stimulation will be 5mA. Heart rate variability during the HFS procedure will be monitored.

After a 25 minutes break the heart rate variability will be assessed a third time during 5 minutes. During the break, subjects will be asked to stay seated, to fill the Pain Catastrophizing scale (short-version) and give a rating from 0-100 for the pain and stress experienced during the HFS procedure (Time7).

Following this break, the area of secondary hyperalgesia will be assessed with a calibrated 128 mN pinprick probe (The Pin Prick, MRC Systems GmbH, Heidelger, Germany) (Time9). Pokes of 1-second duration will be provided at a frequency of 0.5 Hz, starting well outside and approaching the stimulation site with steps of 0,5 cm from 4 different directions towards the application site. Participants will be asked to keep their eyes closed during the entire mapping procedure. Then, participants will rate the pain induced by pin-prick stimulation in the area surrounding the electrode (Time10). This procedure will be conducted three times, with a two-minute break between each assessment (Time 11-14).

The second experimental day (Day2), the procedure will be similar to the first, but informed consent and the Spielberger Trait anxiety inventory and the Pain catastrophization scale will not be filled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* age>18 years and <40 years
* be fluent either in English or French
* ability to provide informed consent

Exclusion Criteria:

* experiencing a pre-existing pain condition
* self-reported medication (except contraceptives) consumption within 48 hours before experimental day and/or self-reported recreational drug use
* presenting any medical conditions, including heart, neurological, dermatological and psychiatric diseases
* participation to more than 6 hours per week of sport
* exhibiting sign of damage at or near the ventral forearm
* tattoos on the tested forearm
* Failure to cooperate to the tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The area of secondary hyperalgesia | 30 minutes (Time9), 35 minutes (Time11) and 40 minutes (Time13) after the application of HFS. There will be two HFS session (Day1 and Day2) separated by at least 15 days. Outcomes are taken at Day1 at Time9, 11 & 13 and on Day 2 at Time9, 11 & 13
  the area of secondary hyperalgesia (cm square) will be assessed with a calibrated 128 mN pinprick probe (The Pin Prick, MRC Systems GmbH, Heidelger, Germany). Pokes of 1-second duration will be provided at a frequency of 0.5 Hz, starting well outside and approaching the stimulation site with steps of 0,5 cm from 4 different directions towards the application site. Participants will be asked to keep their eyes closed during the entire mapping procedure.
Pin-prick pain in the area of secondary hyperalgesia | 5 minutes before (Time2), 33 minutes (Time10), 40 minutes (Time12) and 43 minutes (Time14) after the application of HFS. Outcomes are taken at Day1 at Time2, 10, 12 & 14 and on Day 2 at Time2, 10, 12 & 14
  participants will rate the pain induced by pin-prick stimulation in the area surrounding the electrode on a numerical rating scale ranging from 0 (no perception) to 100 (maximal pain), with 50 representing the transition from nonpainful to painful domains of sensation

SECONDARY OUTCOMES:
Spielberger State Anxiety inventory (total score) | Just before the application of HFS (time 5). Outcome is taken at Day 1 at Time5 and on Day 2 at Time5.
  questionnaire assessing the state of anxiety. The score will range from 20 (low state anxiety) to 80 (high state anxiety).
Spielberger Trait Anxiety inventory (total score) | On day 0, one day before the first testing session (Day 1)
  questionnaire assessing the trait of anxiety. The score will range from 20 (low trait anxiety) to 80 (high trait anxiety). This questionnaire will be sent by email to the participant.
Pain Catastrophization Scale (total score) | On day 0, one day before the first testing session (Day 1)
  questionnaire to assess thoughts and emotions in response to pain. The score will range from 0 (low catastrophization) to 52 (high catastrophization).
Pain catastrophization scale modified version | Just after the application of HFS (time 7). Outcome is taken at Day 1 at Time7 and on Day 2 at Time7.
  questionnaire to assess thoughts and emotions in response to a specific painful event. The score will range from 0 (low catastrophization) to 24 (high catastrophization).
Stress assessment using a Visual Analog Stress scale | Just after the application of HFS (time 7). Outcome is taken at Day 1 at Time 7 and on Day 2 at Time 7.
  Stress on a scale from 0 (low stress) to 100 (maximal stress).
Detection threshold to a single electrical pulse (in mA) | 2 minutes before the application of HFS (Time3). Outcomes are taken at Day1 at Time2 on Day2 at Time2
  Lowest intensity at which the participant feels the electrical pulse
Age | 10 minutes before the application of HFS (Time1). Outcomes are taken at Day1 at Time1 on Day2 at Time1
  Self-declared age of the subject
Size | 10 minutes before the application of HFS (Time1). Outcomes are taken at Day1 at Time1 on Day2 at Time1
  Self-declared size of the subject
Gender | 10 minutes before the application of HFS (Time1). Outcomes are taken at Day1 at Time1 on Day2 at Time1
  Self-declared gender of the subject
Weight | 10 minutes before the application of HFS (Time1). Outcomes are taken at Day1 at Time1 on Day2 at Time1
  Self-declared weight of the subject
Heart rate variability | Continuous assessment from Time1 (10 minutes before the application of HFS) to Time15 (45 minutes after the application of HFS) during each session. Outcome is taken from Time1-Time15 during each of the two testing sessions (Day1 and at Day2)
  changes in the time interval between heart beats through the study completion.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03966508/SAP_000.pdf